CLINICAL TRIAL: NCT01461655
Title: Exploratory Study Evaluating the Efficacy and the Tolerability of the Sequential Application of Two Marketed Products in Patients With Acne Vulgaris, Using a Split-Face Model
Brief Title: Efficacy and the Tolerability of the Sequential Application of Two Marketed Products in Patients With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LP0045-01; 2011-000244-24 (EudraCT Number)
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2016-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical retinoid - Placebo (Placebo Comparator)
  Interventions: Drug: vehicle gel; Drug: marketed topical retinoid
- Topical retinoid-NSAID (Active Comparator)
  Interventions: Drug: marketed topical retinoid; Drug: marketed topical NSAID

INTERVENTIONS:
Drug: marketed topical retinoid — once daily application, 4 weeks
  Arms: Topical retinoid-NSAID
Drug: marketed topical NSAID — once daily application, 4 weeks
  Arms: Topical retinoid-NSAID
Drug: vehicle gel — once daily application, 4 weeks
  Arms: Topical retinoid - Placebo
Drug: marketed topical retinoid — once daily application, 4 weeks
  Arms: Topical retinoid - Placebo

SUMMARY:
The aim of this proof of principle study is to evaluate efficacy and safety of the sequential application of two marketed products for the treatment of acne vulgaris, using the Split-Face model

ELIGIBILITY:
Inclusion Criteria:

* Subjects having understood and signed an informed consent form
* Male or female subjects who are 18 to 35 years (both included) of age presenting acne vulgaris of the face.
* A minimum of 10 inflammatory lesions (papules and pustules) on the entire face, and a minimum of 20 non-inflammatory lesions (open comedones and closed comedones) on the entire face.
* Disease severity grade as mild or moderate according to the investigator's global assessment (grade 2 or grade 3)

Exclusion Criteria:

* Females who are pregnant, of child-bearing potential and who wish to become pregnant during the study, or who are breast feeding.
* Subjects with any acne cysts or more than one nodule per hemiface.
* Subjects with acne conglobata, acne fulminans, secondary acne (e.g. chloracne, drug-induced acne), or any acne requiring systemic treatment.
* Subjects with a dark pigmentation of the skin or skin type that may, in any way, confound interpretation of the study results (skin type V or VI on Fitzpatrick scale.
* Subjects with other facial skin disorders that may interfere with study assessments.
* Subjects who will use medicated cosmetics and/or soaps (including soaps containing antibacterial agents such as benzoyl peroxide, keratolytic agents such as salicylic acid, skin fresheners/astringents or aftershave products) on the face for the duration of the study.
* Subjects with a history of actinic keratosis on the face or skin cancer.
* Use of hormonal oral contraceptives for acne control for less than 6 months prior to the randomisation.
* Subjects using one of the following systemic medication within 4 weeks before the randomisation and during the study, which could have an effect on the trial disease.
* systemic corticosteroids,
* anti-acne drugs,
* oral retinoids
* any immunosuppressive drugs.
* Subjects using systemic NSAIDs (including aspirin) within 1 week before the randomisation and during the study.
* Subjects using paracetamol within 1 week before the randomisation. Paracetamol will be allowed during the study with a maximum dose of 1g twice daily and for a maximum of 3 consecutive days
* Subjects using one of the following topical medication within 2 weeks before the randomisation and during the study, which could have an effect on the trial disease:
* anti-inflammatory drugs (e.g. topical corticosteroids, NSAIDs),
* anti-acne drugs,
* topical retinoids,
* topical antibacterial agents
* any topical immunosuppressive drugs.
* Subjects with known or suspected hypersensitivity to component(s) of the investigational products or other nonsteroidal anti- inflammatory drug NSAIDs (e.g., aspirin, diclofenac, ibuprofen, ketoprofen).
* Subjects with presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting).
* Subjects with known presence of active peptic ulcer.
* Subjects with history (during the last 10 years) or known presence of asthma.
* Subjects with history (during the last 5 years) or known presence of rhinitis or urticaria

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Mrs Queille-Roussel, MD, Principal Investigator — Centre de Pharmacologie Clinique Applique a la Dermatologie
Locations (1):
- CPCAD - Centre de Pharmacologie Clinique Appliquée à la Dermatologie, Nice, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start date: 21-NOV-2011 (FSFV - first subject first visit) Completion date: 26-APR-2012 (LSLV - last subject last visit)
Groups:
- Topical Retinoid - Placebo, Topical Retinoid - NSAID: Using a left-right split face set up, the study evaluated the effect of sequential application of topical retinoid 0.1% gel and NSAID 5% gel in comparison with the sequential application of topical retinoid 0.1% gel and vehicle gel for the treatment of acne vulgaris.
  The randomised subjects received the following products:
  * NSAID 5% gel , in the morning on the appropriate hemiface.
  * Topical retinoid 0.1% gel, in the evening on the entire face.
  * Vehicle gel, in the morning on the appropriate hemiface.
Period: Overall Study
Arm/Group | Topical Retinoid - Placebo, Topical Retinoid - NSAID
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Topical Retinoid - Placebo, Topical Retinoid - NSAID: marketed topical retinoid : once daily application, 4 weeks
  vehicle gel : once daily application, 4 weeks
Arm/Group | Topical Retinoid - Placebo, Topical Retinoid - NSAID
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 17
Region of Enrollment [Number; unit: participants]
  France | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Inflammatory Lesions From Baseline to End of Treatment
Description: Percentage change in inflammatory lesions count from baseline to the end of treatment
Time Frame: Baseline to End of treatment (4 weeks)
Measure: Median (Standard Deviation); unit: percentage of change
Groups:
- Topical Retinoid - Placebo: marketed topical retinoid : once daily application, 4 weeks
  vehicle gel : once daily application, 4 weeks
- Topical Retinoid-NSAID: marketed topical NSAID : once daily application, 4 weeks
  marketed topical retinoid : once daily application, 4 weeks
Arm/Group | Topical Retinoid - Placebo | Topical Retinoid-NSAID
Number analyzed (Participants) | 40 | 40
percentage of change | -20.3 (45.3) | -29.4 (37.0)

2. Secondary Outcome: Non-inflammatory Lesions Count
Description: Percentage change in non-inflammatory lesions count from baseline to the end of treatment
Time Frame: Baseline to End of treatment (4 weeks)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Topical Retinoid - Placebo | Topical Retinoid-NSAID
Number analyzed (Participants) | 40 | 40
percentage of change | -41.4 (31.2) | -43.1 (37.6)

3. Secondary Outcome: Total Lesions Count
Description: Percentage change in total lesions count from baseline to the end of treatment
Time Frame: Baseline to End of treatment (4 weeks)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Topical Retinoid - Placebo | Topical Retinoid-NSAID
Number analyzed (Participants) | 40 | 40
percentage of change | -35.4 (24.0) | -39.9 (27.0)

4. Secondary Outcome: Percentage Change in Total Lesions Count
Description: Percentage change in total leasions count from baseline to day 8
Time Frame: Baseline to Day 8
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Topical Retinoid - Placebo | Topical Retinoid-NSAID
Number analyzed (Participants) | 40 | 40
percentage of change | -20.4 (24.1) | -21.1 (28.6)

5. Secondary Outcome: Percentage Change in Total Lesions Count
Description: Percentage change in total lesions count from baseline to day 15
Time Frame: Baseline to Day 15
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Topical Retinoid - Placebo | Topical Retinoid-NSAID
Number analyzed (Participants) | 40 | 40
percentage of change | -24.9 (24.3) | -22.2 (29.0)

6. Secondary Outcome: Percentage Change in Total Lesions Count
Description: Percentage change in total lesions count from baseline to day 22
Time Frame: Baseline to Day 22
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Topical Retinoid - Placebo | Topical Retinoid-NSAID
Number analyzed (Participants) | 40 | 40
percentage of change | -35.7 (21.8) | -32.5 (30.0)

7. Secondary Outcome: Investigator Global Assessment (IGA) of Disease Severity
Description: The investigator made an assessment of the disease severity (Plaque thickening, Scaling and Erythema) using a 6-point scale (Clear, Almost clear, Mild, Moderate, Severe, and Very severe).
  The outcome was the proportion of "success" (improvement of two grades of the IGA) from baseline to the end of treatment. "Success" is defined as improvement of two grades from the baseline assessment.
Time Frame: Baseline to End of treatment (4 weeks)
Measure: Number; unit: participants
Arm/Group | Topical Retinoid - Placebo | Topical Retinoid-NSAID
Number analyzed (Participants) | 40 | 40
participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study start untill 43 (±2)days after the last on-treatment visit if an AE (serious or non-serious) classified as possible or probably related to the study treatment was ongoing at the last on-treatment visit.
Arm/Group | Topical Retinoid - Placebo, Topical Retinoid - NSAID
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 40/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topical Retinoid - Placebo, Topical Retinoid - NSAID (N=40)
Eyelid oedema (Eye disorders) | 2
Nasopharyngitis (Infections and infestations) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 9
Migraine (Nervous system disorders) | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 7
Eczema (Skin and subcutaneous tissue disorders) | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting or presenting a manuscript, the investigator shall provide to LEO Pharma a copy of all such manuscripts, and LEO Pharma shall have rights to review and comment. Upon the request of LEO Pharma the investigator shall remove any confidential information prior to submitting or presenting the manuscripts. The investigator shall, upon the request of LEO Pharma, delay publication or presentation to allow LEO Pharma to protect its inventions and other intellectual property rights.